CLINICAL TRIAL: NCT01103128
Title: BRCA1 and BRCA2 Genetic Mutations in Mucinous Versus Nonmucinous Precursor Lesions of the Pancreas: Validation of a Mouse Model of Pancreatic Carcinogenesis
Brief Title: Validation of a Mouse Model of Pancreatic Carcinogenesis
Status: Terminated | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Wendy K. Chung, Assistant Professor of Pediatrics, Molecular Genetics, Columbia University
Other Study IDs: AAAE0097; AAAE0097 (Other: Columbia University IRB)
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2012-07

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Pre-neoplastic lesions; Breast and Ovarian Cancer Syndrome; BRCA1/2; Mouse model for pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — * Peripheral Blood Specimens: Three tubes of blood will be collected from each study participant. Two tubes will be EDTA-whole blood and one tube will be serum. Each tube will contain ~4-5 ml. A portion of the blood will be utilized to extract white blood cells that will be immortalized by EBV infection.
  * Archived Fixed Tissue Samples: Tissue blocks from surgery performed at CUMC or elsewhere, will be requested after obtaining consent for study participation.
  * Fresh Tissue Collection: At the time of surgery for tumor resection, tumor and adjacent normal tissue will be requested from the Pathology Department. At the time of endoscopy, aspirated fluid or biopsied tissue will be requested. No additional tissue will be resected beyond that required for surgical or endoscopic management.
  * Genetic Testing: All genetic testing will be performed in a research laboratory. Test results from research laboratories will not be disclosed to patients.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary aim of this study is to determine if mutations of BRCA1 and BRCA2 result in different precancerous pathways to pancreatic ductal adenocarcinoma (PDAC), as suggested in our validated mouse model. Genomic DNA will be isolated on normal tissue obtained from patients who underwent pancreatic resection for PDAC, intraductal papillary mucinous neoplasm (IPMN) or mucinous cystic neoplasm (MCN). Tissue will be examined for the three most common founder mutations in Ashkenazi Jews. In the cases in which BRCA1 or BRCA2 mutations are found, heterozygote normal and abnormal tissue will be examined to look for mutations in the other BRCA1 or BRCA2 allele. The interaction between other cancer causing genes with BRCA1/2 will also be evaluated by comparing the sequences of the other genes in pre-cancerous lesions.

We hypothesize that BRCA1- and BRCA2-mediated pancreatic ductal adenocarcinoma progresses through the PanIN route, as seen in both BRCA1 and BRCA2 murine models of pancreatic cancer. We further hypothesize that BRCA1 mutations may enable an additional pre- neoplastic pathway through MCN, and that IPMN may embody yet another pre- neoplastic pathway.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) is the fourth leading cause of death from malignancy in the United States. Several gene mutations and cancer syndromes have been identified that are found in greater frequency in individuals with PDAC, including the breast ovary cancer syndrome (BRCA1 and BRCA2 mutations). We have recently generated mouse models of pancreatic cancer in which we found that deletions of either BRCA1 or BRCA2 cooperate with K-ras activation and p53 mutations to increase the rate of tumorigenesis via accelerated progression of Pancreatic Intraepithelial Neoplasia (PanIN). However, only BRCA1 deletions were associated with the development of concomitant Mucinous Cystic Neoplasms (MCNs), suggesting potentially distinct pathways for BRCA1- and BRCA2-mediated tumorigenesis in the pancreas. Our primary aim is to determine if germline mutations of BRCA1 and BRCA2 result in different pre-neoplastic pathways to pancreatic cancer, as in our murine model. Genomic DNA will be isolated on normal tissue obtained from patients who underwent pancreatic resection for pancreatic cancer, IPMN or MCN. Tissue will be genotyped for the three most common founder mutations in Ashkenazi Jews. In the cases in which BRCA1 or BRCA2 mutations are found, heterozygote normal and abnormal tissue will be microdissected to look for loss of heterozygosity at the BRCA1 or BRCA2 allele. Our secondary aim is to evaluate the interaction of p53 and Kras with BRCA1 and BRCA2 by sequencing p53 and Kras in PanIN as compared to IPMN and MCN lesions.

ELIGIBILITY:
Inclusion Criteria:

* Tissue-confirmed diagnosis of pancreatic adenocarcinoma, MCN, or IPMN.
* Underwent surgical resection for pancreatic adenocarcinoma, MCN, or IPMN.

Exclusion Criteria:

* Unwilling to provide informed consent.
* Under the age of 18.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects have a tissue-confirmed diagnosis of pancreatic adenocarcinoma, MCN or IPMN and underwent surgical resection for pancreatic adenocarcinoma, MCN or IPMN at Columbia-Presbyterian Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2009-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
BRCA1 vs. BRCA2 mutations | 1 year
  The primary aim is to determine if germline mutations of BRCA1 and BRCA2 result in different pre-neoplastic pathways to pancreatic cancer, as seen in our murine model. Genomic DNA will be isolated on normal tissue obtained from patients who underwent pancreatic resection for pancreatic cancer, IPMN or MCN. Tissue will be genotyped for the three most common founder mutations in Ashkenazi Jews. In the cases in which BRCA1 or BRCA2 mutations are found, heterozygote normal and abnormal tissue will be microdissected to look for loss of heterozygosity at the BRCA1 or BRCA2 allele.

SECONDARY OUTCOMES:
Interaction of other cancer genes with BRCA1 and BRCA2 | 1 year
  The secondary aim is to evaluate the interaction of p53 and K-ras with BRCA1 and BRCA2 by sequencing p53 and K-ras in PanIN as compared to IPMN and MCN lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy K Chung, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States